CLINICAL TRIAL: NCT04927663
Title: A First-in-Human, Phase I PET Imaging Study of 11C-YJH08, a Selective Glucocorticoid Receptor-Targeting Agent, in Patients With Advanced Solid Tumor Malignancies
Brief Title: 11C-YJH08 PET Imaging for Detection of Glucocorticoid Receptor Expression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Rahul Aggarwal (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 20926; NCI-2021-04300 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5R01MH115043-03 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Solid Tumor, Adult; Solid Tumor; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Radioactive Tracers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A: Any Solid Tumor (Dosimetry Cohort) (Experimental): Participants with any solid tumor malignancy with evidence of one or more metastases will receive approximately 20 millicurie (mCi) of 11C-YJH08 IV over 1-2 minutes and 10-60 minutes later, undergo either PET/MRI or PET/CT over 90 minutes at baseline.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: 11C-YJH08; Procedure: Optional Tumor Biopsy
- Cohort B: Metastatic CRPC (Experimental): Participants with metastatic CRPC will receive approximately 20 mCi of 11C-YJH08 IV over 1-2 minutes and 10-60 minutes later, undergo either PET/MRI or PET/CT over 90 minutes at baseline and optional repeat scan at the time of progression.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: 11C-YJH08; Procedure: Optional Tumor Biopsy
- Cohort C: Solid Tumor Malignancy (Experimental): Participants with any solid tumor malignancies other than prostate adenocarcinoma with one or more metastases on conventional imaging will receive approximately 20 mCi of 11C-YJH08 IV over 1-2 minutes and 10-60 minutes later, undergo either PET/MRI or PET/CT over 90 minutes at baseline and optional repeat scan at the time of progression.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: 11C-YJH08; Procedure: Optional Tumor Biopsy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT imaging
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET imaging
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Drug: 11C-YJH08 — Given IV
  Other Names: Radioactive Tag; Radioactive Tracer; Radioactive Label
Procedure: Optional Tumor Biopsy — Optional procedure to obtain tumor tissue
  Other Names: Tumor Biopsy

SUMMARY:
This phase I trial studies if positron emission tomography (PET) imaging using 11C-YJH08 can be useful for detecting certain cell receptor expression in tumor cells in patients with cancer that has spread to other parts of the body (metastatic). 11C-YJH08 is a small-molecule radiotracer that binds to receptors on cells (glucocorticoid receptor) so that they show up better on the PET scan. Systemic therapy (including enzalutamide) can cause more glucocorticoid receptors to be produced in tumor cells, which can make the tumor cells resist hormone therapies. If researchers can find a better way to detect whether glucocorticoid receptors are increasing during therapy, it may lead to more successful therapies using glucocorticoid receptor antagonists.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of metastatic lesion detection in enzalutamide/apalutamide-resistant metastatic castration-resistant prostate cancer (mCRPC) using 11C-YJH08 PET. (Cohort A).

II. To determine the mean percent change from baseline at the time of progression on enzalutamide or apalutamide in standardized uptake value (SUV)max-ave on paired 11C-YJH08 PET on a per-patient and per-lesion basis. (Cohorts B & C).

SECONDARY OBJECTIVES:

I. To determine the safety and determine average organ uptake of 11C-YJH08. II. To descriptively report the patterns of intra-tumoral uptake of 11C-YJH08 on whole body PET, including by site of disease, uptake by tumor type, inter-tumoral and inter-patient heterogeneity, and tumor-to-background signal.

III. To determine whether baseline uptake on 11C-YJH08 PET is associated with subsequent clinical outcomes including objective response rate, progression-free survival, and prostate specific antigen (PSA50) response. (Cohorts B & C)

EXPLORATORY OBJECTIVE:

I. To determine the association between uptake on 11C-YJH08 PET with glucocorticoid receptor (GR) expression and transcriptional signature scores on paired metastatic tumor biopsies.

OUTLINE: Participants are assigned to 1 of 3 arms.

Cohort A (Dosimetry): Participants receive 11C-YJH08 intravenously (IV) over 1-2 minutes and 10-60 minutes later, undergo either PET/magnetic resonance imaging (MRI) or PET/computed tomography (CT) over 90 minutes at baseline.

**Enrollment in Cohorts B & C will enroll after dosimetry has been established in Cohort A**

Cohort B: Participants with mCRPC receive 11C-YJH08 and undergo either PET/MRI or PET/CT at baseline and at time of progression.

Cohort C: Participants with solid tumors receive 11C-YJH08 and undergo either PET/MRI or PET/CT at baseline and at time of progression.

Participants are assessed the day of the scan for safety follow-up, and up to 24 months for non-interventional clinical outcomes. An optional metastatic tumor biopsy may be performed within 14 days of the initial scan.

ELIGIBILITY:
Inclusion Criteria:

1. Disease characteristics by cohort, as defined by:

   * COHORT A: Histologically confirmed metastatic solid tumor malignancy.
   * COHORT B: Metastatic castration-resistant prostate cancer with progression on systemic therapies by Prostate Specific Antigen Working Group 3 (PSAWG3).
   * COHORT C: Metastatic advanced solid tumor malignancy other than prostate adenocarcinoma with at least one metastasis on conventional imaging.
2. The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Age 18 years or older at the time of study entry.
5. Adequate organ function, as defined by:

   1. Serum creatinine =< 1.5 x upper limit of normal (ULN) OR estimated creatinine clearance > 50 ml/min
   2. Total bilirubin =< 1.5 x ULN
   3. Hemoglobin >= 8.0 g/dL
   4. Platelet count >= 50,000/microliter
   5. Absolute neutrophil count >= 1000/microliter

Exclusion Criteria:

1. Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Concurrent treatment with any dose of systemic glucocorticoids within 7 days prior to cycle 1 day 1 (C1D1).
3. History of adrenal insufficiency requiring use of systemic glucocorticoid replacement.
4. History of Cushing's disease or Cushing's syndrome.
5. Any condition that, in the opinion of the principal investigator, would impair the patient's ability to comply with study procedures.
6. Contra-indication to MRI (e.g. pacemaker placement, severe claustrophobia) (applicable only for patients scheduled for PET/MRI).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 2 participants were enrolled to Cohort A. The study was closed for slow accrual before enrollment in Cohort B or Cohort C could begin
Groups:
- Cohort A: Any Solid Tumor (Dosimetry Cohort): Participants with any solid tumor malignancy with evidence of one or more metastases will receive approximately 20 millicurie (mCi) of 11C-YJH08 IV over 1-2 minutes and 10-60 minutes later, undergo either Positron Emission Tomography (PET)/MRI or PET/CT over 90 minutes at baseline.
- Cohort B: Metastatic CRPC: Participants with metastatic castrate resistant prostate cancer (CRPC) will receive approximately 20 mCi of 11C-YJH08 IV over 1-2 minutes and 10-60 minutes later, undergo either PET/MRI or PET/CT over 90 minutes at baseline and optional repeat scan at the time of progression.
Period: Overall Study
Arm/Group | Cohort A: Any Solid Tumor (Dosimetry Cohort) | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study closed before Cohorts B and C could be opened for enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Any Solid Tumor (Dosimetry Cohort) | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Customized [Count of Participants; unit: Participants]
  70-79 years | 1 |  |  | 1
  80-89 years | 1 |  |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  | 0
  Male | 2 |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 1
  Not Hispanic or Latino | 1 |  |  | 1
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of 11C-YJH08 PET in Metastatic Lesion Detection (Cohort A Only)
Description: Using as a cut-off to define a positive lesion on PET as a lesion with SUV at least 1.5 times higher than mediastinal blood pool, the sensitivity (probability that a test will indicate recurrent disease among those with recurrent disease (True Positive / (True Positive + False Negative)) will be descriptively reported on a lesion-per-lesion basis, using as reference standard staging scans including computed tomography or magnetic resonance imaging of the chest/abdomen/pelvis.
Time Frame: Up to day 1 follow-up
Population: Data not collected. Per the pre-specified statistical analysis plan outlined in the study protocol, a sample size of approximately 6 patients for Cohort A is required to collect sufficient data to ensure adequate organ dosimetry and determination of the optimal uptake time following administration of 11C-YJH08.
Arm/Group | Cohort A: Any Solid Tumor (Dosimetry Cohort)
Number analyzed (Participants) | 0

2. Primary Outcome: Median Percent Change From Baseline in Standardized Uptake Value (SUV)Max (Cohort B and C Only)
Description: The median percent change from baseline, and range of SUVmax (across all metastatic lesions per patient) will be descriptively reported using mediastinal blood pool and normal organ as background uptake values.
Time Frame: Up to 24 months
Population: No participants were enrolled in Cohort B or C.
Arm/Group | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Median Percent Change From Baseline at the Time of Progression in Standardized Uptake Value (SUV)Max-ave (Cohort B and C Only)
Description: The median percent change from baseline, and range of SUVmax-ave (in each study cohort) will be descriptively reported using mediastinal blood pool and normal organ as background uptake values.
Time Frame: Up to 24 months
Population: No participants were enrolled in Cohort B or C
Arm/Group | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Reported Treatment-emergent Adverse Events
Description: The frequency and severity of adverse events following 11C-YJH08 injection will be descriptively reported, using NCI Common Terminology Criteria for Adverse Events Version 5.0 criteria.
Time Frame: Up to day 1 after injection
Population: No participants were enrolled in Cohort B or C
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Any Solid Tumor (Dosimetry Cohort) | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 | 0 | 0

5. Secondary Outcome: Median Intra-tumoral Uptake
Description: The median and range for intra-tumoral SUVmax within metastatic lesions will be descriptively reported to asses for intra-tumoral heterogeneity and differences in uptake by site of disease.
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Cohort A: Any Solid Tumor (Dosimetry Cohort) | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Association Between Baseline Uptake on 11C-YJH08 PET With Prostate Specific Antigen (PSA50) Response (Cohort B Only )
Description: The association between baseline and percent change from baseline in SUVmax-ave with the cohort will be dichotomized above and below the median will be compared to the PSA response rate using Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria
Time Frame: Up to 24 months
Population: No participants were enrolled in Cohort B
Arm/Group | Cohort B: Metastatic CRPC
Number analyzed (Participants) | 0

7. Secondary Outcome: Association Between Baseline Uptake on 11C-YJH08 PET and Objective Response Rate (Cohort B & C Only)
Description: The association between baseline and percent change from baseline in SUVmax-ave with the cohort will be dichotomized above and below the median will be compared to the objective response rate (in subset of measurable tumors by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1)
Time Frame: Up to 24 months
Population: No participants were enrolled in Cohort B or C
Arm/Group | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Association Between Baseline Uptake on 11C-YJH08 PET and Clinical Benefit Rate (Cohort B & C Only)
Description: The association between baseline and percent change from baseline in SUVmax-ave with the cohort will be dichotomized above and below the median will be compared to the clinical benefit rate (in subset of measurable tumors by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1)
Time Frame: Up to 24 months
Population: No participants were enrolled in Cohorts B or C
Arm/Group | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Median Progression-free Survival by Cohort (Cohort B & C Only)
Description: The association between baseline and percent change from baseline in SUVmax-ave with the cohort will be dichotomized above and below the median and median progression-free survival will be reported by group.
Time Frame: Up to 24 months
Population: No participants were enrolled in Cohort B or C
Arm/Group | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 days
Description: The study closed to slow accrual before Cohorts B or C could be opened for enrollment.
Arm/Group | Cohort A: Any Solid Tumor (Dosimetry Cohort) | Cohort B: Metastatic CRPC | Cohort C: Solid Tumor Malignancy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study closed earlier than expected due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT04927663/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT04927663/ICF_001.pdf